CLINICAL TRIAL: NCT01613573
Title: A Phase 1, Open-Label, Single and Multiple Dose Study to Assess the Safety and Pharmacokinetics of Pegylated Somatropin(PEG Somatropin) in GHD Children
Brief Title: Crossover Study to Assess the Safety and Pharmacokinetic of Pegylated Somatropin(PEG Somatropin) in GHD Children
Acronym: Phase 1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Changchun GeneScience Pharmaceutical Co., Ltd. (Industry)
Collaborators: Huazhong University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GenSci-004 Clinical Trial
Record Dates: First submitted 2012-06-01; First posted 2012-06-07 (Estimated); Last update posted 2012-06-14 (Estimated); Status verified 2010-10

CONDITIONS: Growth Hormone Deficiency
Keywords: pegylated Somatropin; PEG-GH; Phase 1 study; Pharmacokinetics
MeSH Terms: conditions — Dwarfism, Pituitary | interventions — Human Growth Hormone; Pharmacokinetics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: somatropin AQ — somatropin injection 0.2mg/kg/w once per day, inject for 7 continuous days 4 weeks for cleaning period
  Other Names: Somatropin injection; rhGH
Drug: pegylated somatropin — Pegylated somatropin 0.2mg/kg/w once per week, for continuous 6 weeks Subcutaneous injection
  Other Names: PEG somatropin; PEG GH; pharmacokinetics; growth hormone deficiency

SUMMARY:
The purpose of the phase 1 study is to assess the safety and pharmacokinetics of PEG somatropin, which administered once per week, compared with the daily used somatropin, and to evaluate the safety and possibility to replace daily used somatropin.

ELIGIBILITY:
Inclusion Criteria:

* have a height less than two standard deviations (SD) below the median height for individuals of the same age or height, a growth velocity (GV) ≤4 cm/yr, a GH peak concentration <7 ng/ml in two different provocative tests, a bone age (BA; ≤9 years in girls and ≤10 years in boys) at least 2 years less than his/her chronological age (CA);be in preadolescence (Tanner stage 1) and have a CA >3 years;have a height value recorded 3 months before the start of GH treatment to calculate pre-treatment GV; receive no prior GH treatment or stop the GH treatment for more than 4 weeks;sign informed consent

Exclusion Criteria:

* Patients with Liver and kidney dysfunction (ALT> upper limit of normal 2 times, Cr> upper limit of normal), hepatitis B virus detection, antigen-HBc, HBsAg and HBeAg are positive
* patients with known to a highly allergic constitution or allergic to the drug of this study
* Patients with diabetes, serious cardiopulmonary, blood system, malignant tumor and other diseases or systemic infection in immunocompromised and mental diseases
* Patients with other growth disorders, such as Turner syndrome, constitutional delay of growth and puberty, Laron syndrome, GH receptor deficiency, girls with growth delay have not ruled out chromosomal abnormalities
* Participated in clinical trials of other drugs in 3 months
* Other cases that the researchers considered unsuitable for this clinical trial

Ages: 4 Years to 10 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2010-03; Primary Completion 2010-10 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
pharmacokinetics parameter | Somatropin AQ: predose(0),1,2,3,4,6,8,10,12,16,20,24 hours post-dose. PEG somatropin: predose (0),2,4,8,12,18,24,36,48,72,96,120,144,168 hours post-dose
  Cmax, AUC during the time interval for the first dose and last dose, Half-Life(t1/2), Apparent body clearance(CL), Mean residence time(MRT),steady-state volume of distribution(Vss)

SECONDARY OUTCOMES:
IGF-1, IGFBP-3 | Day I to Day 7 in each treatment period (33 time points) for daily used somatropin, Day I to Day 42 in each treatment period (35 time points) for PEG somatropin

CONTACTS AND LOCATIONS:
Overall Officials: Luo Xiaoping, Doctor, Principal Investigator — Tongji Hospital